CLINICAL TRIAL: NCT03034967
Title: Randomised, Double-Blind (Sponsor Open), Placebo-Controlled, Multicentre, Dose Ranging Study to Evaluate the Efficacy and Safety of Danirixin Tablets Administered Twice Daily Compared With Placebo for 24 Weeks in Adult Participants With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Danirixin Dose Ranging Study in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205724; 2016-003675-21 (EudraCT Number)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: HCRU exacerbations; SGRQ; CXCR2 antagonist; GSK1325756; Danirixin; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Danirixin 5 mg (Experimental): Eligible participants will receive danirixin 5 mg tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin; Drug: Standard of care; Drug: Rescue medication
- Danirixin 10 mg (Experimental): Eligible participants will receive danirixin 10 mg tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin; Drug: Standard of care; Drug: Rescue medication
- Danirixin 25 mg (Experimental): Eligible participants will receive danirixin 25 mg tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin; Drug: Standard of care; Drug: Rescue medication
- Danirixin 35 mg (Experimental): Eligible participants will receive danirixin 35 mg tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin; Drug: Standard of care; Drug: Rescue medication
- Danirixin 50 mg (Experimental): Eligible participants will receive danirixin 50 mg tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin; Drug: Standard of care; Drug: Rescue medication
- Placebo (Placebo Comparator): Eligible participants will receive placebo tablet with food twice daily along with standard care of treatment for 24 weeks.
  Interventions: Drug: Danirixin matching placebo; Drug: Standard of care; Drug: Rescue medication

INTERVENTIONS:
Drug: Danirixin — Danirixin is available as 5, 10, 25, 35 and 50 mg white, film-coated, oval or round shaped tablets for oral administration.
  Arms: Danirixin 10 mg; Danirixin 25 mg; Danirixin 35 mg; Danirixin 5 mg; Danirixin 50 mg
Drug: Danirixin matching placebo — Danirixin matching placebo will be available as white, film-coated, oval or round shaped tablets for oral administration.
  Arms: Placebo
Drug: Standard of care — Participants will continue with their standard of care inhaled medications (i.e. long acting bronchodilators with or without inhaled corticosteroids) during the study treatment.
Drug: Rescue medication — Participants will continue to use rescue medication(s). The following rescue medications may be used: short acting beta agonists, short acting muscarinic antagonists, or short acting combination bronchodilators.

SUMMARY:
Danirixin (DNX) is a selective CXC chemokine receptor (CXCR2) antagonist being developed as a potential anti-inflammatory agent for the treatment of COPD. This is a Phase 2, randomized, double-blind (Sponsor Open) study. The primary objective of the study is to evaluate the clinical activity and safety of danirixin compared with placebo in participants with COPD. Following baseline assessments collected over a 7 day period participants will be randomized (1:1:1:1:1:1) to receive one of five dose strengths of danirixin (5 milligram [mg], 10 mg, 25 mg, 35 mg and 50 mg) or placebo. Study treatment will be administered orally twice daily for 24 weeks. Participants will continue with their standard of care inhaled medications (i.e. long acting bronchodilators with or without inhaled corticosteroids) while receiving study treatment. Follow up will continue up to 28 days post last dose. Approximately 700 participants will be screened with a target of 540 participants completing 24 weeks of treatment and key study assessments.

ELIGIBILITY:
Inclusion Criteria

* Participants must be aged between 40 to 80 years of age inclusive, at the time of signing the informed consent.
* Participants who have COPD (post bronchodilator FEV1/FVC ratio <0.7 and FEV1% predicted >=40%) based on American Thoracic Society (ATS)/European Respiratory Society (ERS) current guidelines. Participants with a historical diagnosis of asthma may be included so long as they have a current diagnosis of COPD.
* History of respiratory symptoms including chronic cough, mucus hypersecretion, and dyspnea on most days for at least the previous 3 months prior to screening.
* Participants with a documented history of COPD exacerbation(s) in the 12 months prior to study participation (screening) meeting at least one of the following criteria: >=2 COPD exacerbations resulting in prescription for antibiotics and/or oral corticosteroids or hospitalization or extended observation in a hospital emergency room or outpatient center; 1 COPD exacerbation resulting in prescription for antibiotics and/or oral corticosteroids of hospitalization or extended observation in a hospital emergency room or outpatient center and a plasma fibrinogen concentration at screening >=3 grams/liter (300 milligram/deciliter)
* Current and former smokers with a cigarette smoking history of >=10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or equivalent). Current smokers are defined as those who are currently smoking cigarettes (i.e. have smoked at least one cigarette daily or most days for the month prior to Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Participants must have the ability and willingness to use an electronic diary (log pad) on a daily basis.
* Body weight >=45 kilogram (kg)
* Male or female: A male participant must agree to use contraception during the treatment period and for at least 60 hours after the last dose of study treatment, corresponding to approximately 6 half-lives (which is the time needed to eliminate any teratogenic study treatment) and to refrain from donating sperm during this period; A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 60 hours after the last dose of study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria

* Diagnosis of other clinically relevant lung diseases (other than COPD), e.g. sarcoidosis, tuberculosis, pulmonary fibrosis, severe bronchiectasis or lung cancer.
* Alpha-1-antitrypsin deficiency as the underlying cause of COPD
* Pulse oximetry <88% at rest at screening. Participants should be tested while breathing room air. However, participants living at high altitudes (above 5000 feet or 1500 meters above sea level) who are receiving supplemental oxygen can be included provided they are receiving the equivalent of <4 liter per minute (L/min) and screening pulse oximetry is measured while on their usual oxygen settings.
* Less than 14 days have elapsed from the completion of a course of antibiotics or oral corticosteroids for a recent COPD exacerbation.
* A peripheral blood neutrophil count <1.5 x 10^9/L.
* Diagnosis of pneumonia (chest X-ray or CT confirmed) within the 3 months prior to screening.
* Chest x-ray (posterior-anterior with lateral) or CT scan reveals evidence of a clinically significant abnormality not believed to be due to the presence of COPD (historic results up to 1 year prior to screening may be used). For sites in Germany: If a chest x-ray (or CT scan) within 1 year prior to screening is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office of Radiation Protection (BfS).
* History or current evidence of other clinically significant medical condition that is uncontrolled on permitted therapies. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through study participation, or that would affect the safety analysis or other analysis if the disease/condition worsened during the study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Abnormal and clinically significant 12-lead ECG finding. The investigator will determine the clinical significance of each abnormal ECG finding in relation to the participant's medical history and exclude participants who would be at undue risk by participating in the study. An abnormal and clinically significant finding that would preclude a participant from entering the study is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: atrial fibrillation with rapid ventricular rate >120 beats per minute (bpm); sustained or non-sustained ventricular tachycardia; second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator has been implanted); Corrected QT Interval using Fridericia formula (QTcF) >=500 millisecond (msec) in participants with QRS <120 msec and QTcF >=530 msec in participants with QRS >=120 msec.
* Previous lung surgery (e.g. lobectomy, pneumonectomy) or lung volume reduction procedure.
* Current or expected chronic use of macrolide antibiotics during the study period for the prevention of COPD exacerbations. Examples of chronic use include, but are not limited to, daily or two to three times per week use for at least 3 months.
* Oral or injectable CYP3A4 or breast cancer resistance protein (BRCP) substrates with a narrow therapeutic index (CYP3A4 substrates include, but are not limited to, alfenatil, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, and theophylline; BRCP substrates include, but are not limited to, topotecan.) The Investigator should consult with the Medical Monitor if necessary.
* Current or expected use of phosphodiesterase-4 inhibitors (e.g. roflumilast). Participants currently receiving roflumilast may be included if they are able to discontinue use from 30 days prior to screening through the completion of the follow up visit.
* Participation in a previous clinical trial and has received an investigational product within any of the following time periods prior to the first dosing day in the current study: 30 days, 5 half lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in a previous clinical trial with danirixin within 1 year prior to the first dosing day in the current study
* Exposure to more than four investigational products within 1 year prior to the first dosing day in the current study.
* Alanine transferase (ALT) >2x upper limit of normal (ULN); bilirubin > 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* A positive test for human immunodeficiency virus (HIV) antibody
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result within 3 months prior to screening.
* Pulmonary rehabilitation: Participants who have taken part in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to screening or participants who plan to enter the acute phase of a pulmonary rehabilitation program during the study. Participants who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* A history of allergy or hypersensitivity to any of the ingredients in the study treatment.
* A known or suspected history of alcohol or drug abuse within the 2 years prior to screening.
* Inability to read: in the opinion of the Investigator, any participant who is unable to read and/or would not be able to complete study related materials.
* Affiliation with the study site: study investigators, sub-investigators, study coordinators, employees of a study investigator, sub-investigator or study site, or immediate family member of any of the above that are involved with the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- United States (8):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Morgantown, West Virginia
- Australia (5):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
- Canada (6):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- Germany (7):
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Netherlands (5):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
- Poland (5):
  - GSK Investigational Site, Ksawerów
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Wroclaw
- Romania (9):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Focşani
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Slobozia
  - GSK Investigational Site, Suceava
- South Korea (4):
  - GSK Investigational Site, Bucheon-Si, Gyeonggi-Do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wonju-si, Gangwon-do
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20593

REFERENCES:
- [Background] Lazaar AL, Miller BE, Donald AC, Keeley T, Ambery C, Russell J, Watz H, Tal-Singer R; for 205724 Investigators. CXCR2 antagonist for patients with chronic obstructive pulmonary disease with chronic mucus hypersecretion: a phase 2b trial. Respir Res. 2020 Jun 12;21(1):149. doi: 10.1186/s12931-020-01401-4. PMID 32532258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the dose response and safety of danirixin compared with placebo in Chronic Obstructive Pulmonary Disease (COPD) participants with respiratory symptoms including cough, increased sputum production and dyspnoea.
Pre-assignment Details: A total of 614 participants were randomized in this study across 9 countries.
Groups:
- Placebo: Participants received placebo film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
- Danirixin 5 mg: Participants received danirixin 5 milligram (mg) film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
- Danirixin 10 mg: Participants received danirixin 10 mg film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
- Danirixin 25 mg: Participants received danirixin 25 mg film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
- Danirixin 35 mg: Participants received danirixin 35 mg film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
- Danirixin 50 mg: Participants received danirixin 50 mg film coated tablets orally twice daily with food and standard care of treatment for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Started | 102 | 102 | 103 | 103 | 102 | 102
Completed | 88 | 97 | 90 | 92 | 88 | 87
Not Completed | 14 | 5 | 13 | 11 | 14 | 15
Not completed — Withdrawal by Subject | 9 | 2 | 6 | 6 | 9 | 2
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Liver function test abnormality | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 2 | 1 | 1 | 0
Not completed — Adverse Event, non-fatal | 3 | 1 | 2 | 0 | 2 | 8
Not completed — Adverse Event, Serious Fatal | 0 | 1 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg | Total
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102 | 614
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (7.31) | 66.3 (6.79) | 65.7 (7.48) | 66.3 (7.28) | 65.1 (7.58) | 65.7 (6.98) | 65.9 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 32 | 38 | 35 | 32 | 202
  Male | 73 | 66 | 71 | 65 | 67 | 70 | 412
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 10 | 6 | 18 | 17 | 10 | 17 | 78
  Asian - South East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 1 | 0 | 0 | 1 | 6
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White - Arabic/North African Heritage | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White - White/Caucasian/European Heritage | 87 | 93 | 84 | 86 | 92 | 84 | 526

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Respiratory Symptoms Measured by Evaluating Respiratory Symptoms (E-RS) in COPD. E-RS: COPD Total Score
Description: E-RS: COPD is a subset of Exacerbations of Chronic pulmonary Disease Tool (EXACT). E-RS is a tool that consists of 11 items from the 14 item EXACT instrument. The domains include: respiratory symptoms (RS)-breathlessness (RS-BRL comprised of 5 items, score range [0-17]), RS-cough and sputum (RS-CSP comprised of 3 items, score range [0-11]), and RS-chest symptoms (RS-CSY comprised of 3 items, score range [0-12]). The total score ranged between 0-40 and higher values indicates severe respiratory symptoms. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Per protocol population included all participants from the mITT population who did not have a protocol deviation considered to impact efficacy. Posterior mean change and standard deviation has been presented.
Time Frame: Baseline and Month 6
Population: Per Protocol Population. Only those participants with data available at the specified data points was analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 86 | 95 | 87 | 91 | 85 | 86
Scores on a scale | -2.11 (0.345) | -1.93 (0.289) | -1.47 (0.349) | -0.87 (0.286) | -0.76 (0.259) | -0.71 (0.281)
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.08, 90% CI 2-sided [0.00 to 0.66] — Median posterior difference, 90 percent (%) credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; 4-parameter Emax model; Test type: Other — Emax; Median Posterior Difference = 0.61, 90% CI 2-sided [0.00 to 1.52] — Median posterior difference, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 1.25, 90% CI 2-sided [0.43 to 1.97] — Median posterior difference, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 1.34, 90% CI 2-sided [0.72 to 2.03] — Median posterior difference, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 1.38, 90% CI 2-sided [0.79 to 2.07] — Median posterior difference, 90% credible interval for Placebo and Danirixin 50 mg has been presented

2. Primary Outcome: Change From Baseline in Respiratory Symptoms Measured by E-RS in COPD (E-RS: COPD Breathlessness Score)
Description: E-RS: COPD is a subset of EXACT. E-RS is a tool that consists of 11 items from the 14 item EXACT instrument. The domains include: RS-BRL comprised of 5 items, score range (0-17), RS-CSP comprised of 3 items, score range (0-11), and RS-CSY comprised of 3 items, score range (0-12). The total score ranged between 0-40 and higher values indicates severe respiratory symptoms. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Posterior mean change and standard deviation has been presented.
Time Frame: Baseline and Month 6
Population: Per Protocol Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 86 | 95 | 87 | 91 | 85 | 86
Scores on a scale | -0.82 (0.202) | -0.69 (0.162) | -0.41 (0.183) | -0.15 (0.148) | -0.10 (0.141) | -0.09 (0.158)
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.09, 90% CI 2-sided [0.00 to 0.42] — Median posterior difference, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; 4-parameter Emax model; Test type: Other — Emax; Median Posterior Difference = 0.43, 90% CI 2-sided [0.00 to 0.87] — Median posterior difference, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.68, 90% CI 2-sided [0.23 to 1.08] — Median posterior difference, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.72, 90% CI 2-sided [0.37 to 1.10] — Median posterior difference, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.73, 90% CI 2-sided [0.40 to 1.12] — Median posterior difference, 90% credible interval for Placebo and Danirixin 50 mg has been presented

3. Primary Outcome: Change From Baseline in Respiratory Symptoms Measured by E-RS in COPD (E-RS: COPD Cough and Sputum Score)
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: Per Protocol Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 86 | 95 | 87 | 91 | 85 | 86
Scores on a scale | -0.83 (0.107) | -0.79 (0.090) | -0.67 (0.109) | -0.46 (0.104) | -0.40 (0.088) | -0.37 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.01, 90% CI 2-sided [0.00 to 0.16] — Median posterior difference, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; 4-parameter Emax model; Test type: Other — Emax; Median Posterior Difference = 0.12, 90% CI 2-sided [0.00 to 0.43] — Median posterior difference, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.38, 90% CI 2-sided [0.04 to 0.61] — Median posterior difference, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.42, 90% CI 2-sided [0.21 to 0.64] — Median posterior difference, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; 4-parameter Emax model selected; Test type: Other — Emax; Median Posterior Difference = 0.45, 90% CI 2-sided [0.26 to 0.66] — Median posterior difference, 90% credible interval for Placebo and Danirixin 50 mg has been presented

4. Primary Outcome: Change From Baseline in Respiratory Symptoms Measured by E-RS in COPD (E-RS: COPD Chest Symptoms Score)
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: Per Protocol Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 86 | 95 | 87 | 91 | 85 | 86
Scores on a scale | -0.36 (0.148) | -0.35 (0.061) | -0.34 (0.062) | -0.34 (0.069) | -0.34 (0.073) | -0.34 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Log-linear model; Test type: Other — Log-linear; Median Posterior Difference = 0.01, 90% CI 2-sided [-0.21 to 0.23] — Median posterior difference, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Log-linear model; Test type: Other — Log-linear; Median Posterior Difference = 0.01, 90% CI 2-sided [-0.23 to 0.25] — Median posterior difference, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Log-linear model; Test type: Other — Log-linear; Median Posterior Difference = 0.01, 90% CI 2-sided [-0.27 to 0.29] — Median posterior difference, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Log-linear model; Test type: Other — Log-linear; Median Posterior Difference = 0.01, 90% CI 2-sided [-0.28 to 0.30] — Median posterior difference, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Log-linear model; Test type: Other — Log-linear; Median Posterior Difference = 0.01, 90% CI 2-sided [-0.29 to 0.31] — Median posterior difference, 90% credible interval for Placebo and Danirixin 50 mg has been presented

5. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Time Frame: Up to Day 196
Population: Modified Intent-to-Treat (mITT) population. mIIT population comprised of all randomized participants who were randomized apart from those randomized in error, received a treatment randomization number, modified and data for this population were based on actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Participants
  Any AE | 63 | 63 | 69 | 68 | 63 | 71
  Any SAE | 8 | 7 | 13 | 10 | 7 | 11

6. Primary Outcome: Number of Participants With Worst Case Hematology Parameter Results by Potential Clinical Importance (PCI)
Description: Blood samples were collected from participants for analysis of following hematology parameters with PCI low and high values: Basophils % (High 5.00x), Eosinophils % (High 2.00x), Mean corpuscular hemoglobin concentration (MCHC) gram per deciliter (g/dL) (Low 0.85x, high 1.10x), Mean corpuscular hemoglobin (MCH) picograms (pg) (Low 0.85x, high 1.20x), Mean corpuscular volume (MCV) femtoliter (fL) (low 0.25x, high 2.00x), Erythrocytes (Ery.)(10^12cells/L) (Low 0.93x, high 1.07x), Hematocrit (Ratio of 1) (Low 0.50x, high 0.50x), Hemoglobin gram per liter (g/L) (Low 0.85x, high 1.20x), Leukocytes (x10^9/L) (Low 0.70x, high 1.60x), Lymphocytes % (Low 0.80x, high 1.20x), Monocytes % (Low 0.80x, high 1.60x), Neutrophils % (Low 0.65x, high 1.50x), Platelets (x10^9cells/L) (Low 0.90x, high 1.10x). Multipliers are identified by "x", otherwise actual comparison values are provided with units. Values above and below this range were considered of PCI.
Time Frame: Up to Day 196
Population: mITT population. Only those participants with available data at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Participants
  Basophils, No change, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Basophils, No change, n=97, 102, 101, 101, 101, 99 | 97 | 102 | 101 | 101 | 101 | 99
  Basophils, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Basophils, High, n=97, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils,No change,n=97,102,101,101,101,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Eosinophils,No change,n=97,102,101,101,101,99 | 97 | 101 | 101 | 98 | 100 | 98
  Eosinophils, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Eosinophils, High, n=97, 102, 101, 101, 101, 99 | 0 | 1 | 0 | 3 | 1 | 1
  Ery. MCHC, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCHC, Low, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. MCHC,No change,n=97,102,101,101,102,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCHC,No change,n=97,102,101,101,102,99 | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCHC, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCHC, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. MCH, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCH, Low, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 1
  Ery. MCH, No Change, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCH, No Change, n=97, 102, 101, 101, 102, 99 | 97 | 102 | 101 | 101 | 102 | 98
  Ery. MCH, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCH, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. MCV, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCV, Low, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. MCV, No Change, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCV, No Change, n=97, 102, 101, 101, 102, 99 | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCV, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Ery. MCV, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Erythrocytes, Low, n=97, 102, 101, 101, 102, 99 | 2 | 1 | 3 | 3 | 2 | 2
  Erythrocytes, No change,n=97,102,101,101,102,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Erythrocytes, No change,n=97,102,101,101,102,99 | 93 | 99 | 97 | 97 | 99 | 97
  Erythrocytes. High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Erythrocytes. High, n=97, 102, 101, 101, 102, 99 | 2 | 2 | 1 | 1 | 1 | 0
  Hematocrit, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hematocrit, Low, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, No Change, n=97,102,101,101,102,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hematocrit, No Change, n=97,102,101,101,102,99 | 97 | 102 | 101 | 101 | 102 | 99
  Hematocrit, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hematocrit, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hemoglobin, Low, n=97, 102, 101, 101, 102, 99 | 1 | 1 | 2 | 0 | 2 | 0
  Hemoglobin, No change, n=97,102,101,101,102,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hemoglobin, No change, n=97,102,101,101,102,99 | 96 | 101 | 99 | 101 | 100 | 99
  Hemoglobin, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Hemoglobin, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, Low, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Leukocytes, Low, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocytes, No change, n=97,102,101,101,102,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Leukocytes, No change, n=97,102,101,101,102,99 | 97 | 102 | 101 | 101 | 102 | 98
  Leukocytes, High, n=97, 102, 101, 101, 102, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 102 | 99
  Leukocytes, High, n=97, 102, 101, 101, 102, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Low, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Lymphocytes, Low, n=97, 102, 101, 101, 101, 99 | 3 | 7 | 5 | 8 | 7 | 4
  Lymphocytes, No change, n=97,102,101,101,101,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Lymphocytes, No change, n=97,102,101,101,101,99 | 94 | 95 | 96 | 92 | 93 | 94
  Lymphocytes, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Lymphocytes, High, n=97, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 1 | 1 | 1
  Monocytes, No change, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Monocytes, No change, n=97, 102, 101, 101, 101, 99 | 97 | 101 | 99 | 101 | 100 | 98
  Monocytes, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Monocytes, High, n=97, 102, 101, 101, 101, 99 | 0 | 1 | 2 | 0 | 1 | 1
  Neutrophils, Low, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Neutrophils, Low, n=97, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 1 | 3 | 1
  Neutrophils, No change, n=97,102,101,101,101,99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Neutrophils, No change, n=97,102,101,101,101,99 | 97 | 102 | 101 | 100 | 98 | 98
  Neutrophils, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Neutrophils, High, n=97, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, Low, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Platelets, Low, n=97, 102, 101, 101, 101, 99 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets, No change, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Platelets, No change, n=97, 102, 101, 101, 101, 99 | 97 | 99 | 100 | 101 | 99 | 99
  Platelets, High, n=97, 102, 101, 101, 101, 99: number analyzed (Participants) | 97 | 102 | 101 | 101 | 101 | 99
  Platelets, High, n=97, 102, 101, 101, 101, 99 | 0 | 2 | 1 | 0 | 2 | 0

7. Primary Outcome: Number of Participants With Worst Case Clinical Chemistry Parameter Results by PCI
Description: Blood samples were collected from participants for analysis of following chemistry parameters with PCI low and high values: Alanine aminotransferase (ALT) International units per liter (IU/L) (High => 3x ULN), Alkaline phosphatase (ALP) (IU/L) (High ≥ 2x ULN); Aspartate aminotransferase (AST) (IU/L) (High=> 3x ULN); Bilirubin micromole per liter (umol/L) (High ≥ 2x ULN); Calcium millimole per liter (mmol/L) (Low 0.85x, high 1.08x), Chloride (mmol/L) (Low 0.90x, high 1.10x), Creatinine (umol/L) (High 1.30x), Direct bilirubin (umol/L) (High ≥ 2x ULN), Glucose (mmol/L) (Low <0.6x, high >4x), Potassium (mmol/L) (Low 0.75x, high 1.30x); Protein (g/L) (High 1.25x), Sodium (mmol/L) (Low 0.80x, high 1.15x), Multipliers are identified by "x", otherwise actual comparison values are provided with units. Values above and below this range were considered of PCI.
Time Frame: Up to Day 196
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Participants
  ALT, No change,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  ALT, No change,n=99,102,102,102,101,100 | 99 | 102 | 101 | 102 | 101 | 100
  ALT, High, n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  ALT, High, n=99,102,102,102,101,100 | 0 | 0 | 1 | 0 | 0 | 0
  ALP, No change,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  ALP, No change,n=99,102,102,102,101,100 | 99 | 102 | 102 | 102 | 101 | 100
  ALP, High, n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  ALP, High, n=99,102,102,102,101,100 | 0 | 0 | 0 | 0 | 0 | 0
  AST, No change,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  AST, No change,n=99,102,102,102,101,100 | 99 | 102 | 101 | 102 | 101 | 100
  AST, High, n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  AST, High, n=99,102,102,102,101,100 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin, No change, n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Bilirubin, No change, n=99,102,102,102,101,100 | 99 | 101 | 102 | 102 | 101 | 100
  Bilirubin, High, n=99, 102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Bilirubin, High, n=99, 102,102,102,101,100 | 0 | 1 | 0 | 0 | 0 | 0
  Calcium, Low, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Calcium, Low, n=96,102,101,101,101,99 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, No change, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Calcium, No change, n=96,102,101,101,101,99 | 96 | 102 | 101 | 101 | 101 | 99
  Calcium, High, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Calcium, High, n=96,102,101,101,101,99 | 0 | 0 | 0 | 0 | 0 | 0
  CO2, Low, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  CO2, Low, n=96,102,101,101,101,99 | 1 | 0 | 2 | 1 | 0 | 1
  CO2, No change, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  CO2, No change, n=96,102,101,101,101,99 | 94 | 102 | 99 | 99 | 101 | 98
  CO2, High, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  CO2, High, n=96,102,101,101,101,99 | 1 | 0 | 0 | 1 | 0 | 0
  Chloride, Low, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Chloride, Low, n=96,102,101,101,101,99 | 0 | 0 | 0 | 0 | 0 | 0
  Chloride, No change, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Chloride, No change, n=96,102,101,101,101,99 | 96 | 102 | 101 | 101 | 101 | 99
  Chloride, High, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Chloride, High, n=96,102,101,101,101,99 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, No change, n=96,102,101,101,101,99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Creatinine, No change, n=96,102,101,101,101,99 | 94 | 100 | 99 | 99 | 99 | 99
  Creatinine, High, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Creatinine, High, n=96, 102, 101, 101, 101, 99 | 2 | 2 | 2 | 2 | 2 | 0
  Direct bilirubin,NoChange,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Direct bilirubin,NoChange,n=99,102,102,102,101,100 | 98 | 102 | 102 | 102 | 101 | 100
  Direct bilirubin,High,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Direct bilirubin,High,n=99,102,102,102,101,100 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose, Low, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Glucose, Low, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, No change, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Glucose, No change, n=96, 102, 101, 101, 101, 99 | 96 | 102 | 101 | 101 | 101 | 99
  Glucose, High, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Glucose, High, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, Low, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Potassium, Low, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, No change, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Potassium, No change, n=96, 102, 101, 101, 101, 99 | 96 | 102 | 101 | 101 | 101 | 99
  Potassium, High, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Potassium, High, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Protein, No change, n=99, 102, 102, 102, 101, 100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Protein, No change, n=99, 102, 102, 102, 101, 100 | 99 | 102 | 102 | 102 | 101 | 100
  Protein, High, n=99, 102, 102, 102, 101, 100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Protein, High, n=99, 102, 102, 102, 101, 100 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, Low, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Sodium, Low, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, No change, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Sodium, No change, n=96, 102, 101, 101, 101, 99 | 96 | 102 | 101 | 101 | 101 | 99
  Sodium, High, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Sodium, High, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Urea, Low, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Urea, Low, n=96, 102, 101, 101, 101, 99 | 0 | 0 | 0 | 0 | 0 | 0
  Urea, No change, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Urea, No change, n=96, 102, 101, 101, 101, 99 | 96 | 101 | 101 | 100 | 101 | 98
  Urea, High, n=96, 102, 101, 101, 101, 99: number analyzed (Participants) | 96 | 102 | 101 | 101 | 101 | 99
  Urea, High, n=96, 102, 101, 101, 101, 99 | 0 | 1 | 0 | 1 | 0 | 1
  Bilirubin/ALT,No change,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Bilirubin/ALT,No change,n=99,102,102,102,101,100 | 99 | 102 | 102 | 102 | 101 | 100
  Bilirubin/ALT, High,n=99,102,102,102,101,100: number analyzed (Participants) | 99 | 102 | 102 | 102 | 101 | 100
  Bilirubin/ALT, High,n=99,102,102,102,101,100 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Worst Case Vital Signs Parameter Results by PCI
Description: Vital signs parameters includes systolic blood pressure (SBP) and diastolic blood pressure (DBP), pulse rate and respiration rate were measured in a semi-supine position after 5 minutes rest for the participants at indicated time points. PCI ranges for vital signs parameters were as follows: <90 to >160 millimeters of mercury (mmHg) for SBP and <40 to >110 mmHg for DBP, <35 or >120 beats per minute for heart rate and <8 or >30 breaths per minute for respiration rate. Values above and below this range were considered of PCI.
Time Frame: Up to Day 168
Population: mITT population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 96 | 102 | 101 | 101 | 102 | 99
Participants
  SBP, Low | 0 | 0 | 0 | 0 | 0 | 1
  SBP, No change | 93 | 92 | 95 | 98 | 98 | 94
  SBP, High | 3 | 10 | 6 | 3 | 4 | 4
  DBP, Low | 0 | 0 | 0 | 0 | 0 | 0
  DBP, No change | 96 | 102 | 101 | 101 | 102 | 99
  DBP, High | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, Low | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, No change | 96 | 102 | 99 | 100 | 102 | 98
  Pulse rate, High | 0 | 0 | 2 | 1 | 0 | 1
  Respiratory rate, Low | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory rate, No change | 96 | 102 | 101 | 101 | 102 | 98
  Respiratory rate, High | 0 | 0 | 0 | 0 | 0 | 1

9. Primary Outcome: Number of Participants With Worst Case Post-Baseline Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECG obtained to measure PR, QRS, QT, and Corrected QT intervals. Only those participants with worst case post-Baseline data have been represented for abnormal - not clinical significant and abnormal - clinical significant. Day 1 was considered as Baseline.
Time Frame: Baseline and Day 168
Population: mITT population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 96 | 102 | 101 | 101 | 102 | 99
Participants
  Not Clinical significant | 52 | 65 | 68 | 67 | 62 | 53
  Clinical significant | 2 | 1 | 1 | 0 | 3 | 1

10. Secondary Outcome: Number of Moderate or Severe Healthcare Resource Utilization (HCRU) Exacerbations Per Participant
Description: Participants with moderate or severe COPD exacerbations, i.e. breathlessness, cough, sputum production, chest congestion and chest tightness analyzed. Mild exacerbations are defined as exacerbations that did not require treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization, Emergency Room [ER] visit or resulting in death). Moderate exacerbations are defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization, ER visit or resulting in death). Severe exacerbations are defined as exacerbations that required hospitalization, ER visit or resulted in death. Number of moderate or severe HCRU exacerbations per participant has been presented, where 0= participants in each treatment group who did not experience an event; 1= participants in each treatment group who experienced 1 event and >=2= participants in each treatment group who experienced 2 or more events.
Time Frame: Up to Day 196
Population: Per Protocol Population.
Measure: Number; unit: Exacerbations per participant
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Exacerbations per participant
  0 | 66 | 51 | 61 | 63 | 55 | 50
  1 | 28 | 34 | 23 | 28 | 30 | 36
  >=2 | 7 | 17 | 16 | 12 | 15 | 13

11. Secondary Outcome: Number of Responders E-RS in COPD (E-RS): COPD Total Score
Description: E-RS: COPD is a subset of EXACT. E-RS is a tool that consists of 11 items from the 14 item EXACT instrument. E-RS is intended to capture information related to the respiratory symptoms of COPD, i.e. breathlessness, cough, sputum production, chest congestion and chest tightness. The E-RS has a scoring range of 0-40; higher scores indicate more severe symptoms. Response is defined as an E-RS: COPD total score of 2 units below baseline or lower. Non-response is defined as an E-RS: COPD total score higher than 2 units below Baseline.
Time Frame: Month 6
Population: Per Protocol Population. Number of participants presented represent those with data available at the time point being presented; however, all participants in the per protocol population without missing covariate information and with at least one post baseline measurement are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 86 | 95 | 87 | 91 | 85 | 86
Participants | 33 | 48 | 33 | 30 | 29 | 32
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other; p = 0.089, linear mixed model — Analysis performed using a generalized linear mixed model with a logit link function including treatment, relevant Baseline E-RS: COPD score, smoking status at Screening, country, month, Baseline by month and treatment by month interactions; Odds Ratio (OR) = 1.71, 90% CI 2-sided [1.02 to 2.86] — Odds Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other; p = 0.881, linear mixed model — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.05, 90% CI 2-sided [0.62 to 1.79] — Odds Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other; p = 0.674, linear mixed model — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.87, 90% CI 2-sided [0.51 to 1.48] — Odds Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other; p = 0.804, linear mixed model — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.92, 90% CI 2-sided [0.54 to 1.58] — Odds Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other; p = 0.987, linear mixed model — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.01, 90% CI 2-sided [0.59 to 1.71] — Odds Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented

12. Secondary Outcome: Number of EXACT Events Per Participant
Description: EXACT is a 14 item patient reported outcome (PRO) instrument designed to capture information on the occurrence, frequency, severity, and duration of exacerbations of disease in participants with COPD. The total score for EXACT-PRO ranges from 0-100, higher scores indicate more severe symptoms. Events were categorized as recovered, censored, or persistent worsening. Number of EXACT events per participant has been presented, where 0= participants in each treatment group who did not experience an event; 1= participants in each treatment group who experienced 1 event and >=2= participants in each treatment group who experienced 2 or more events.
Time Frame: Up to Day 196
Population: Per Protocol Population.
Measure: Number; unit: Events
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Events
  0 | 92 | 92 | 92 | 92 | 86 | 86
  1 | 9 | 6 | 7 | 9 | 10 | 10
  >=2 | 0 | 4 | 1 | 2 | 4 | 3

13. Secondary Outcome: Time to First EXACT Event
Description: The time to first on-treatment EXACT event was calculated as the onset date of the first on-treatment EXACT event minus date of start of treatment plus 1.
Time Frame: Up to Day 168
Population: Per Protocol Population.
Measure: Number; unit: Days
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Days
  First quartile (Q1) time to event | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment.
  Median time to event | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment.
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other; Median Posterior Hazard Ratio = 1.2, 90% CI 2-sided [0.5 to 2.6] — Median Posterior Hazard Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented; DNX versus (vs.) Placebo statistics calculated using a Bayesian proportional hazards model including treatment, gender, exacerbation history (<=1/>=2 moderate/severe), smoking status at Screening, country and post-bronchodilator % predicted Forced Expiratory Volume in one second (FEV1)at Screening
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other; Median Posterior Hazard Ratio = 1.0, 90% CI 2-sided [0.4 to 2.4] — Median Posterior Hazard Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented; DNX vs. Placebo statistics calculated using a Bayesian proportional hazards model including treatment, gender, exacerbation history (<=1/>=2 moderate/severe), smoking status at Screening, country and post-bronchodilator % predicted FEV1 at Screening
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other; Median Posterior Hazard Ratio = 1.4, 90% CI 2-sided [0.6 to 3.2] — Median Posterior Hazard Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other; Median Posterior Hazard Ratio = 2.0, 90% CI 2-sided [1.0 to 4.3] — Median Posterior Hazard Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other; Median Posterior Hazard Ratio = 2.0, 90% CI 2-sided [0.9 to 4.5] — Median Posterior Hazard Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented; [other analysis details as in outcome 13, analysis 2]

14. Secondary Outcome: Severity of EXACT Event
Description: EXACT is a 14 item PRO instrument designed to capture information on the occurrence, frequency, severity, and duration of exacerbations of disease in participants with COPD. The total score for EXACT-PRO ranges from 0-100, higher scores indicate more severe symptoms. Severity is the highest EXACT total score during the period from onset to recovery.
Time Frame: Up to Day 168
Population: Per Protocol Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 9 | 15 | 9 | 13 | 19 | 16
Scores on a scale | 22.1 (6.60) | 26.7 (3.71) | 22.9 (5.28) | 28.6 (5.68) | 25.0 (5.54) | 26.4 (6.36)

15. Secondary Outcome: EXACT Event Duration for All Events
Description: EXACT is a 14 item PRO instrument designed to capture information on the occurrence, frequency, severity, and duration of exacerbations of disease in participants with COPD. The total score for EXACT-PRO ranges from 0-100, higher scores indicate more severe symptoms. Severity is the highest EXACT total score during the period from onset to recovery. Duration of EXACT events has been reported.
Time Frame: Up to Day 168
Population: Per Protocol Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 9 | 15 | 9 | 13 | 19 | 16
Days | 45.3 (50.37) | 11.6 (10.15) | 45.8 (51.97) | 25.5 (42.11) | 17.6 (16.28) | 18.7 (37.75)

16. Secondary Outcome: Time to First HCRU-defined COPD Exacerbation
Description: The time to first on-treatment Moderate/Severe HCRU exacerbation was calculated as exacerbation onset date of first on-treatment moderate or severe on-treatment exacerbation - date of start of treatment +1.
Time Frame: Up to Day 196
Population: Per Protocol Population.
Measure: Number; unit: Days
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Days
  Q1 time to event | 110 | 47 | 63 | 79 | 70 | 57
  Median time to event | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | 152
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.5, 90% CI 2-sided [1.0 to 2.2] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented; DNX vs. Placebo statistics calculated using a Bayesian proportional hazards model including treatment, gender, exacerbation history (<=1/>=2 moderate/severe), smoking status at Screening, country and post-bronchodilator %predicted FEV1 at Screening
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.1, 90% CI 2-sided [0.8 to 1.7] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.1, 90% CI 2-sided [0.7 to 1.6] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.4, 90% CI 2-sided [1.0 to 2.1] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.6, 90% CI 2-sided [1.1 to 2.3] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented; [other analysis details as in outcome 13, analysis 2]

17. Secondary Outcome: Time to First Severe HCRU-defined COPD Exacerbation
Description: A COPD exacerbation defined as a severe exacerbation if it requires hospitalization or ER visit or extended observation. The time to first on-treatment Moderate/Severe HCRU exacerbation was calculated as exacerbation onset date of first on-treatment moderate or severe on-treatment exacerbation - date of start of treatment +1.
Time Frame: Up to Day 196
Population: Per Protocol Population.
Measure: Number; unit: Days
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Days
  Q1 time to event | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment. | NA — If <25% of participants experienced the event within a treatment then Q1 time to event are displayed as NA (not applicable) for that treatment.
  Median time to event | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment. | NA — If <50% of participants experienced the event within a treatment then median time to event are displayed as NA (not applicable) for that treatment.
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.8, 90% CI 2-sided [0.7 to 5.5] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.9, 90% CI 2-sided [0.7 to 5.8] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 1.8, 90% CI 2-sided [0.7 to 5.6] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 2.3, 90% CI 2-sided [0.9 to 6.9] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented; [other analysis details as in outcome 13, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other — Bayesian proportional hazards model; Hazard Ratio (HR) = 0.8, 90% CI 2-sided [0.2 to 2.7] — Hazard Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented; [other analysis details as in outcome 13, analysis 2]

18. Secondary Outcome: HCRU-defined Exacerbation Duration
Description: The duration of HCRU exacerbation were determined. The duration of the exacerbation was calculated as (exacerbation resolution date or date of death - exacerbation onset date + 1). For exacerbations which were not resolved but where the participant later died from other causes, the duration was calculated using date of death as the end date of the event.
Time Frame: Up to Day 196
Population: Per Protocol Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 44 | 75 | 58 | 56 | 66 | 65
Days | 10.3 (7.37) | 12.3 (8.95) | 12.9 (9.58) | 14.0 (8.71) | 10.7 (7.21) | 14.2 (9.29)

19. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Total Score
Description: The SGRQ-C consists of 40 items aggregated into 3 component scores: Symptoms, Activity, Impacts, and a Total score. Each response to a question is assigned a weight. Component scores are calculated by summing the weights from all positive items in that component, dividing by the sum of weights for all items in that component, and multiplying this number by 100. Component scores could range from 0-100, with a higher component score indicating greater disease burden. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Posterior mean change and standard deviation has been presented.
Time Frame: Baseline, Days 84 and 168
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Scores on a scale
  Day 84, n=93, 97, 94, 96, 91, 90: number analyzed (Participants) | 93 | 97 | 94 | 96 | 91 | 90
  Day 84, n=93, 97, 94, 96, 91, 90 | -3.79 (1.172) | -3.63 (1.150) | -1.31 (1.146) | -3.19 (1.148) | -2.83 (1.189) | -2.48 (1.175)
  Day 168, n=85, 96, 86, 90, 86, 85: number analyzed (Participants) | 85 | 96 | 86 | 90 | 86 | 85
  Day 168, n=85, 96, 86, 90, 86, 85 | -4.11 (1.292) | -3.44 (1.246) | -4.19 (1.292) | -4.94 (1.251) | -4.12 (1.287) | -3.41 (1.302)

20. Secondary Outcome: Number of SGRQ Responder
Description: A participant was consider Responder according to SGRQ total score if their change from Baseline SGRQ total score of 4 units below Baseline or lower.
Time Frame: Day 84 and Day 168
Population: Per Protocol Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Participants
  Day 84, n=93, 97, 94, 96, 91, 90: number analyzed (Participants) | 93 | 97 | 94 | 96 | 91 | 90
  Day 84, n=93, 97, 94, 96, 91, 90 | 39 | 40 | 35 | 49 | 35 | 38
  Day 168, n=85, 96, 86, 90, 86, 85: number analyzed (Participants) | 85 | 96 | 86 | 90 | 86 | 85
  Day 168, n=85, 96, 86, 90, 86, 85 | 35 | 47 | 40 | 47 | 41 | 34
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other; p = 0.208, Linear mixed model — Analysis performed using a generalized linear mixed model with a logit link function including treatment, Baseline SGRQ total score, smoking status at Screening, country, visit, Baseline by visit and treatment by visit interactions; Odds Ratio (OR) = 1.51, 90% CI 2-sided [0.88 to 2.59] — Odds Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other; p = 0.482, Linear mixed model — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 1.27, 90% CI 2-sided [0.73 to 2.20] — Odds Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other; p = 0.239, Linear mixed model — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 1.47, 90% CI 2-sided [0.86 to 2.53] — Odds Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other; p = 0.426, Linear mixed model — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 1.31, 90% CI 2-sided [0.75 to 2.26] — Odds Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other; p = 0.763, Linear mixed model — [p-value comment as in outcome 20, analysis 1]; Odds Ratio (OR) = 0.90, 90% CI 2-sided [0.52 to 1.58] — Odds Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented

21. Secondary Outcome: Change From Baseline COPD Assessment Test (CAT) Total Score
Description: The CAT is an 8 item questionnaire (cough, sputum, chest tightness, breathlessness, going up hills/stairs, activity limitation at home, confidence leaving the home, and sleep and energy) that measures health status of participants with COPD. Participants were completed each question by rating their experience on a 6 point scale ranging from 0 (maximum impairment) to 5 (no impairment) with a total scoring range of 0-40; higher scores indicate worse health status. A CAT score was calculated by summing the non-missing scores on the eight items. Individual items are scored from 0 to 5 with a total score range from 0 - 40, higher scores indicate greater disease impact. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Posterior mean change and standard deviation has been presented.
Time Frame: Baseline, Days 84 and 168
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Scores on a scale
  Day 84, n=89, 97, 92, 89, 88, 85: number analyzed (Participants) | 89 | 97 | 92 | 89 | 88 | 85
  Day 84, n=89, 97, 92, 89, 88, 85 | -2.02 (0.536) | -0.86 (0.525) | -0.63 (0.524) | -0.55 (0.542) | -1.51 (0.543) | -0.36 (0.549)
  Day 168, n=84, 94, 86, 87, 85, 83: number analyzed (Participants) | 84 | 94 | 86 | 87 | 85 | 83
  Day 168, n=84, 94, 86, 87, 85, 83 | -1.39 (0.557) | -1.39 (0.537) | -1.23 (0.548) | -0.97 (0.560) | -1.56 (0.560) | -1.32 (0.565)

22. Secondary Outcome: Number of CAT Responder
Description: A participant was considered as a responder according to CAT score if their change from Baseline CAT score 2.0 units below Baseline or lower.
Time Frame: Day 84 and Day 168
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Participants
  Day 84, n=89, 97, 92, 89, 88, 85: number analyzed (Participants) | 89 | 97 | 92 | 89 | 88 | 85
  Day 84, n=89, 97, 92, 89, 88, 85 | 46 | 44 | 38 | 37 | 43 | 36
  Day 168, n=84, 94, 86, 87, 85, 83: number analyzed (Participants) | 84 | 94 | 86 | 87 | 85 | 83
  Day 168, n=84, 94, 86, 87, 85, 83 | 41 | 44 | 39 | 42 | 46 | 44
Statistical Analysis 1: Comparison: Placebo vs Danirixin 5 mg; Test type: Other; p = 0.973, Linear mixed model — Analysis performed using a generalized linear mixed model with a logit link function including treatment, Baseline CAT score, smoking status at Screening, country, visit, Baseline by visit and treatment by visit interactions; Odds Ratio (OR) = 1.01, 90% CI 2-sided [0.58 to 1.76] — Odds Ratio, 90% credible interval for Placebo and Danirixin 5 mg has been presented
Statistical Analysis 2: Comparison: Placebo vs Danirixin 10 mg; Test type: Other; p = 0.825, Linear mixed model — [p-value comment as in outcome 22, analysis 1]; Odds Ratio (OR) = 0.93, 90% CI 2-sided [0.53 to 1.63] — Odds Ratio, 90% credible interval for Placebo and Danirixin 10 mg has been presented
Statistical Analysis 3: Comparison: Placebo vs Danirixin 25 mg; Test type: Other; p = 0.887, Linear mixed model — [p-value comment as in outcome 22, analysis 1]; Odds Ratio (OR) = 0.95, 90% CI 2-sided [0.55 to 1.66] — Odds Ratio, 90% credible interval for Placebo and Danirixin 25 mg has been presented
Statistical Analysis 4: Comparison: Placebo vs Danirixin 35 mg; Test type: Other; p = 0.567, Linear mixed model — [p-value comment as in outcome 22, analysis 1]; Odds Ratio (OR) = 1.21, 90% CI 2-sided [0.69 to 2.13] — Odds Ratio, 90% credible interval for Placebo and Danirixin 35 mg has been presented
Statistical Analysis 5: Comparison: Placebo vs Danirixin 50 mg; Test type: Other; p = 0.501, Linear mixed model — [p-value comment as in outcome 22, analysis 1]; Odds Ratio (OR) = 1.26, 90% CI 2-sided [0.72 to 2.20] — Odds Ratio, 90% credible interval for Placebo and Danirixin 50 mg has been presented

23. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 as a Lung Function Assessment
Description: Spirometric analysis was done to determine FEV1. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Least square mean change from Baseline and standard error has been presented.
Time Frame: Baseline, Days 84 and 168
Population: mITT Population. Number of participants presented represent those with data available at the time point being presented; however, all participants in the mITT population without missing covariate information and with at least one post baseline measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Liters
  Day 84, n=94, 99, 98, 97, 92, 93: number analyzed (Participants) | 94 | 99 | 98 | 97 | 92 | 93
  Day 84, n=94, 99, 98, 97, 92, 93 | 0.016 (0.0208) | -0.031 (0.0203) | -0.029 (0.0204) | -0.018 (0.0206) | -0.027 (0.0211) | 0.027 (0.0210)
  Day 168, n=88, 97, 90, 90, 88, 86: number analyzed (Participants) | 88 | 97 | 90 | 90 | 88 | 86
  Day 168, n=88, 97, 90, 90, 88, 86 | -0.016 (0.0199) | -0.043 (0.0191) | -0.033 (0.0197) | -0.058 (0.0198) | -0.012 (0.0201) | -0.011 (0.0202)

24. Secondary Outcome: Percent Predicted Normal FEV1
Description: Spirometric analysis was done to determine percent predicted FEVI at screening. FEV1 is forced expiratory volume in one second. Percent predicted FEV1 is defined as the percent FEV1 of the participant is divided by average FEV1 percent in the population of any person similar age, sex and body composition.
Time Frame: At Screening
Population: Per Protocol Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 100 | 102 | 100 | 103 | 100 | 99
Percent predicted FEV1 | 58.98 (12.838) | 56.75 (12.038) | 56.62 (11.848) | 56.84 (12.813) | 57.51 (14.076) | 57.84 (12.794)

25. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Vital Capacity (FVC) as a Lung Function Assessment
Description: Spirometric analysis was done to determine FVC. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Least square mean change from Baseline and standard error has been presented.
Time Frame: Baseline, Days 84 and 168
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Liters
  Day 84, n=94, 99, 98, 97, 92, 93: number analyzed (Participants) | 94 | 99 | 98 | 97 | 92 | 93
  Day 84, n=94, 99, 98, 97, 92, 93 | 0.024 (0.0321) | -0.054 (0.0313) | -0.043 (0.0315) | 0.027 (0.0317) | -0.049 (0.0326) | 0.014 (0.0323)
  Day 168, n=88, 97, 90, 90, 88, 86: number analyzed (Participants) | 88 | 97 | 90 | 90 | 88 | 86
  Day 168, n=88, 97, 90, 90, 88, 86 | -0.011 (0.0348) | -0.079 (0.0335) | -0.043 (0.0344) | -0.024 (0.0345) | -0.036 (0.0351) | -0.016 (0.0353)

26. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1/FVC Ratio as a Lung Function Assessment
Description: Spirometric analysis was done to determine FEV1 and FVC. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Days 84 and 168
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Ratio of FEV1/FVC
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102
Ratio of FEV1/FVC
  Day 84, n=94, 99, 98, 97, 92, 93: number analyzed (Participants) | 94 | 99 | 98 | 97 | 92 | 93
  Day 84, n=94, 99, 98, 97, 92, 93 | -0.003 (0.0543) | -0.001 (0.0554) | -0.000 (0.0453) | -0.013 (0.0630) | -0.000 (0.0402) | 0.014 (0.1636)
  Day 168, n=88, 97, 90, 90, 88, 86: number analyzed (Participants) | 88 | 97 | 90 | 90 | 88 | 86
  Day 168, n=88, 97, 90, 90, 88, 86 | -0.007 (0.0622) | -0.003 (0.0555) | 0.003 (0.0420) | -0.015 (0.0610) | 0.002 (0.0495) | -0.002 (0.0385)

27. Secondary Outcome: Change From Baseline Number of Puffs of Rescue Medication Per Day
Description: The mean number of puffs of rescue per day was calculated over the same time periods and using the same assumptions as rescue use via diary. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Least square mean change from Baseline and standard error has been presented.
Time Frame: Baseline, Months 1, 2, 3, 4, 5 and 6
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Puffs per day
  Month 1, n=100, 102, 100, 102, 98, 99: number analyzed (Participants) | 100 | 102 | 100 | 102 | 98 | 99
  Month 1, n=100, 102, 100, 102, 98, 99 | 0.00 (0.132) | 0.36 (0.130) | 0.28 (0.132) | 0.15 (0.130) | -0.03 (0.133) | 0.28 (0.133)
  Month 2, n=96, 100, 98, 97, 98, 96: number analyzed (Participants) | 96 | 100 | 98 | 97 | 98 | 96
  Month 2, n=96, 100, 98, 97, 98, 96 | -0.22 (0.187) | 0.42 (0.184) | 0.18 (0.186) | 0.35 (0.185) | 0.07 (0.187) | 0.33 (0.188)
  Month 3, n=95, 100, 95, 97, 94, 92: number analyzed (Participants) | 95 | 100 | 95 | 97 | 94 | 92
  Month 3, n=95, 100, 95, 97, 94, 92 | -0.18 (0.184) | 0.29 (0.181) | 0.21 (0.184) | 0.25 (0.182) | 0.07 (0.185) | 0.27 (0.186)
  Month 4, n=92, 98, 92, 97, 90, 90: number analyzed (Participants) | 92 | 98 | 92 | 97 | 90 | 90
  Month 4, n=92, 98, 92, 97, 90, 90 | -0.18 (0.193) | 0.27 (0.189) | 0.27 (0.192) | 0.21 (0.190) | -0.04 (0.194) | 0.44 (0.195)
  Month 5, n=88, 97, 88, 94, 87, 87: number analyzed (Participants) | 88 | 97 | 88 | 94 | 87 | 87
  Month 5, n=88, 97, 88, 94, 87, 87 | -0.16 (0.190) | 0.17 (0.186) | 0.19 (0.190) | 0.25 (0.187) | -0.06 (0.191) | 0.29 (0.192)
  Month 6, n=86, 95, 88, 91, 85, 86: number analyzed (Participants) | 86 | 95 | 88 | 91 | 85 | 86
  Month 6, n=86, 95, 88, 91, 85, 86 | -0.17 (0.196) | 0.21 (0.191) | 0.10 (0.195) | 0.15 (0.193) | 0.04 (0.197) | 0.28 (0.198)

28. Secondary Outcome: Participant Experience of Physical Activity Measured Using PROactive Physical Activity in COPD (C-PPAC) Questionnaire
Description: The Clinical Visit PROactive Physical Activity in COPD (C-PPAC) tool is a designed for intermittent use within a clinical study. PROactive Total Score and two domain scores (amount and difficulty) are derived using data from the C-PPAC questionnaire and a physical activity monitor worn for 7 days prior to the questionnaire.C-PPAC is a 12 item questionnaire. The PROactive tools are scored from 0 to 100 with higher scores indicating greater disease impact. It was implemented in a subset of approximately 50% of participants. The amount domain is calculated using 2 items from the C-PPAC questionnaire (amount of walking outside and chores outside) and 2 activity monitor outputs (vector magnitude units per minute (VMU/min) and steps/day). Each domain score is based on the addition of items (0-15 for amount and 0-40 for difficulty) and then scaled from 0-100. The total score is calculated as (amount+difficulty)/2.
Time Frame: Days 84 and 168
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 101 | 102 | 100 | 103 | 100 | 99
Scores on a scale
  Total score, Day 84, n=8, 4, 6, 6, 10, 6: number analyzed (Participants) | 8 | 4 | 6 | 6 | 10 | 6
  Total score, Day 84, n=8, 4, 6, 6, 10, 6 | 3.00 (5.964) | -5.75 (6.035) | -3.83 (12.754) | 0.42 (2.635) | -1.20 (8.453) | 2.33 (2.677)
  Total score, Day 168, n=13, 7, 9, 8, 6, 7: number analyzed (Participants) | 13 | 7 | 9 | 8 | 6 | 7
  Total score, Day 168, n=13, 7, 9, 8, 6, 7 | -0.96 (13.266) | 1.86 (9.344) | 2.11 (5.878) | 1.25 (3.423) | 4.08 (6.492) | 0.43 (7.607)
  Amount score, Day 84, n=8, 4, 6, 6, 10, 6: number analyzed (Participants) | 8 | 4 | 6 | 6 | 10 | 6
  Amount score, Day 84, n=8, 4, 6, 6, 10, 6 | 2.25 (5.825) | -8.50 (7.937) | -4.00 (19.204) | 0.00 (6.957) | -4.20 (10.706) | -0.83 (5.345)
  Amount score, Day 168, n=13, 7, 9, 8, 6, 7: number analyzed (Participants) | 13 | 7 | 9 | 8 | 6 | 7
  Amount score, Day 168, n=13, 7, 9, 8, 6, 7 | -3.69 (14.733) | -0.43 (8.810) | 2.11 (9.558) | 1.25 (9.161) | 3.67 (11.708) | -4.14 (12.522)
  Difficult score, Day 84, n=29, 22, 18, 19, 24, 14: number analyzed (Participants) | 29 | 22 | 18 | 19 | 24 | 14
  Difficult score, Day 84, n=29, 22, 18, 19, 24, 14 | 6.38 (9.511) | 1.64 (8.301) | -0.17 (7.679) | 1.89 (11.704) | 2.79 (9.278) | 4.50 (9.598)
  Difficult score, Day 168, n=29, 20, 18, 19, 25, 15: number analyzed (Participants) | 29 | 20 | 18 | 19 | 25 | 15
  Difficult score, Day 168, n=29, 20, 18, 19, 25, 15 | 3.03 (14.409) | 2.20 (11.039) | 2.11 (7.553) | 0.63 (11.413) | 1.52 (9.687) | 4.87 (8.887)

29. Secondary Outcome: Danirixin Whole Blood Pharmacokinetic Concentration-Time Data
Description: Blood samples were collected from the participants for the analysis of blood pharmacokinetic concentration-time data. All participants in the mITT population who had at least 1 non-missing Pharmacokinetic assessment obtained and analyzed whilst on treatment with danirixin were included Pharmacokinetic population.
Time Frame: Pre-dose on Days 1, 56, 84 and 168; 0.5, 1, 2, 4, 6, 8, 10, 12 hours post-dose on Days 1 and 168
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 103 | 102 | 102 | 101
Nanogram per milliliter
  Day 1, Pre-dose, n=97, 99, 102, 102, 100: number analyzed (Participants) | 97 | 99 | 102 | 102 | 100
  Day 1, Pre-dose, n=97, 99, 102, 102, 100 | 2.1 (19.41) | 0.4 (3.92) | 0.3 (3.06) | 17.2 (169.33) | 3.9 (39.10)
  Day 1, 0.5 hour, n=16, 19, 24, 26, 19: number analyzed (Participants) | 16 | 19 | 24 | 26 | 19
  Day 1, 0.5 hour, n=16, 19, 24, 26, 19 | 86.7 (85.73) | 210.4 (207.54) | 730.5 (1046.42) | 976.1 (839.37) | 1331.0 (1220.06)
  Day 1, 1 hour, n=16, 18, 24, 26, 19: number analyzed (Participants) | 16 | 18 | 24 | 26 | 19
  Day 1, 1 hour, n=16, 18, 24, 26, 19 | 148.3 (104.75) | 343.3 (228.66) | 822.0 (527.47) | 1183.5 (760.02) | 1846.2 (979.95)
  Day 1, 2 hours, n=16, 19, 24, 26, 19: number analyzed (Participants) | 16 | 19 | 24 | 26 | 19
  Day 1, 2 hours, n=16, 19, 24, 26, 19 | 115.3 (46.00) | 277.7 (245.32) | 707.7 (256.63) | 1011.2 (398.82) | 1472.8 (858.49)
  Day 1, 4 hours, n=16, 19, 24, 26, 19: number analyzed (Participants) | 16 | 19 | 24 | 26 | 19
  Day 1, 4 hours, n=16, 19, 24, 26, 19 | 59.2 (17.79) | 165.3 (136.50) | 401.5 (188.75) | 591.5 (302.96) | 904.6 (599.85)
  Day 1, 6 hours, n=16, 19, 24, 26, 19: number analyzed (Participants) | 16 | 19 | 24 | 26 | 19
  Day 1, 6 hours, n=16, 19, 24, 26, 19 | 34.4 (12.32) | 100.6 (84.26) | 270.0 (169.37) | 371.5 (335.23) | 594.9 (525.00)
  Day 1, 8 hours, n=15, 19, 24, 26, 19: number analyzed (Participants) | 15 | 19 | 24 | 26 | 19
  Day 1, 8 hours, n=15, 19, 24, 26, 19 | 26.1 (13.54) | 67.8 (61.02) | 213.8 (162.24) | 325.8 (359.79) | 428.2 (398.16)
  Day 1, 10 hours, n=16, 18, 22, 26, 19: number analyzed (Participants) | 16 | 18 | 22 | 26 | 19
  Day 1, 10 hours, n=16, 18, 22, 26, 19 | 42.5 (67.85) | 61.5 (56.67) | 265.0 (396.25) | 274.5 (328.04) | 302.3 (255.81)
  Day 1, 12 hours, n=16, 16, 21, 26, 18: number analyzed (Participants) | 16 | 16 | 21 | 26 | 18
  Day 1, 12 hours, n=16, 16, 21, 26, 18 | 87.2 (174.14) | 74.7 (82.51) | 188.2 (188.27) | 232.8 (316.67) | 459.3 (561.53)
  Day 56, Pre-dose, n=94, 91, 94, 95, 92: number analyzed (Participants) | 94 | 91 | 94 | 95 | 92
  Day 56, Pre-dose, n=94, 91, 94, 95, 92 | 53.2 (73.19) | 91.8 (102.43) | 252.3 (295.15) | 372.1 (427.41) | 572.0 (738.28)
  Day 84, Pre-dose, n=97, 94, 96, 91, 90: number analyzed (Participants) | 97 | 94 | 96 | 91 | 90
  Day 84, Pre-dose, n=97, 94, 96, 91, 90 | 50.2 (77.78) | 76.2 (106.86) | 212.3 (211.35) | 342.8 (411.28) | 484.3 (527.47)
  Day 168, Pre-dose, n=92, 85, 89, 85, 84: number analyzed (Participants) | 92 | 85 | 89 | 85 | 84
  Day 168, Pre-dose, n=92, 85, 89, 85, 84 | 41.2 (38.02) | 99.5 (138.00) | 217.9 (221.92) | 350.7 (336.07) | 459.5 (421.30)
  Day 168, 0.5 hours, n=14, 12, 17, 18, 16: number analyzed (Participants) | 14 | 12 | 17 | 18 | 16
  Day 168, 0.5 hours, n=14, 12, 17, 18, 16 | 147.7 (91.51) | 248.3 (189.30) | 530.5 (536.75) | 1449.5 (949.00) | 1635.6 (1077.48)
  Day 168, 1 hours, n=14, 13, 17, 18, 16: number analyzed (Participants) | 14 | 13 | 17 | 18 | 16
  Day 168, 1 hours, n=14, 13, 17, 18, 16 | 162.1 (108.88) | 314.0 (157.04) | 681.2 (630.86) | 1590.3 (1019.32) | 1725.4 (870.79)
  Day 168, 2 hours, n=14, 13, 17, 18, 16: number analyzed (Participants) | 14 | 13 | 17 | 18 | 16
  Day 168, 2 hours, n=14, 13, 17, 18, 16 | 127.4 (88.80) | 331.9 (164.10) | 574.7 (445.85) | 1045.2 (414.21) | 1736.6 (592.51)
  Day 168, 4 hours, n=13, 11, 16, 18, 16: number analyzed (Participants) | 13 | 11 | 16 | 18 | 16
  Day 168, 4 hours, n=13, 11, 16, 18, 16 | 90.5 (53.67) | 190.9 (103.35) | 452.8 (289.44) | 805.0 (346.87) | 1459.9 (909.32)
  Day 168, 6 hours, n=13, 13, 16, 18, 15: number analyzed (Participants) | 13 | 13 | 16 | 18 | 15
  Day 168, 6 hours, n=13, 13, 16, 18, 15 | 55.6 (26.36) | 135.5 (87.39) | 289.6 (188.04) | 554.8 (313.52) | 960.4 (633.37)
  Day 168, 8 hours, n=13, 13, 17, 18, 15: number analyzed (Participants) | 13 | 13 | 17 | 18 | 15
  Day 168, 8 hours, n=13, 13, 17, 18, 15 | 41.5 (19.75) | 102.6 (60.14) | 245.1 (165.40) | 444.9 (298.69) | 760.8 (679.30)
  Day 168, 10 hours, n=13, 12, 17, 18, 15: number analyzed (Participants) | 13 | 12 | 17 | 18 | 15
  Day 168, 10 hours, n=13, 12, 17, 18, 15 | 42.4 (35.98) | 76.6 (56.95) | 193.9 (128.42) | 380.2 (285.81) | 715.0 (840.54)
  Day 168, 12 hours, n=13, 12, 17, 18, 15: number analyzed (Participants) | 13 | 12 | 17 | 18 | 15
  Day 168, 12 hours, n=13, 12, 17, 18, 15 | 42.2 (41.29) | 73.1 (41.21) | 169.7 (114.20) | 481.2 (640.17) | 662.4 (877.91)

30. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Time of Quantifiable Concentration [AUC(0-t)] of Danirixin in Whole Blood Using Dried Blood Spot
Description: Blood samples were collected at indicated timepoints for the analysis of phamacokinetic parameter. All participants in the PK population who had at least 1 non-missing PK assessment obtained and analyzed whilst on treatment with danirixin from a dry blood spot sample and corresponding wet whole blood sample were included in Pharmacokinetic population.
Time Frame: Days 1 and 168
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*nanogram per milliliter
Arm/Group | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 103 | 102 | 102 | 101
Hour*nanogram per milliliter
  Day 1, n=17, 19, 24, 26, 19: number analyzed (Participants) | 17 | 19 | 24 | 26 | 19
  Day 1, n=17, 19, 24, 26, 19 | 543.0 [354.9 to 830.8] | 1373.1 [1081.7 to 1743.0] | 3851.5 [3136.7 to 4729.2] | 5485.1 [4604.8 to 6533.8] | 8073.4 [6591.3 to 9888.7]
  Day 168, n=14, 13, 17, 18, 16: number analyzed (Participants) | 14 | 13 | 17 | 18 | 16
  Day 168, n=14, 13, 17, 18, 16 | 752.1 [546.8 to 1034.4] | 1701.8 [1257.2 to 2303.7] | 4170.1 [3198.1 to 5437.6] | 7682.6 [6384.8 to 9244.0] | 11538.0 [9313.4 to 14294.0]

31. Secondary Outcome: Concentration Maximum (Cmax) of Danirixin in Whole Blood Using Dried Blood Spots
Description: Blood samples were collected from the participants for the analysis of pharmacokinetic parameter.
Time Frame: Days 1 and 168
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter
Arm/Group | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 103 | 102 | 102 | 101
Nanogram per milliliter
  Day 1, n=17, 19, 24, 26, 19: number analyzed (Participants) | 17 | 19 | 24 | 26 | 19
  Day 1, n=17, 19, 24, 26, 19 | 164.9 [119.5 to 227.5] | 343.1 [264.1 to 445.6] | 1028.8 [818.2 to 1293.7] | 1386.2 [1172.1 to 1639.3] | 2119.1 [1728.9 to 2597.4]
  Day 168, n=14, 13, 17, 18, 16: number analyzed (Participants) | 14 | 13 | 17 | 18 | 16
  Day 168, n=14, 13, 17, 18, 16 | 171.9 [123.5 to 239.4] | 357.3 [274.4 to 465.4] | 821.2 [570.9 to 1181.2] | 1695.0 [1285.8 to 2234.5] | 2390.5 [2014.6 to 2836.5]

32. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Danirixin in Whole Blood Using Dried Blood Spots
Description: Blood samples were collected from the participants for the analysis of pharmacokinetic parameter.
Time Frame: Days 1 and 168
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
Number analyzed (Participants) | 102 | 103 | 102 | 102 | 101
Hours
  Day 1, n=17, 19, 24, 26, 19: number analyzed (Participants) | 17 | 19 | 24 | 26 | 19
  Day 1, n=17, 19, 24, 26, 19 | 1.000 [0.58 to 11.80] | 1.000 [0.50 to 12.00] | 1.000 [0.50 to 10.08] | 1.000 [0.48 to 5.85] | 1.000 [0.50 to 12.00]
  Day 168, n=14, 13, 17, 18, 16: number analyzed (Participants) | 14 | 13 | 17 | 18 | 16
  Day 168, n=14, 13, 17, 18, 16 | 1.000 [0.50 to 11.78] | 1.000 [0.50 to 2.00] | 1.000 [0.33 to 10.00] | 1.000 [0.48 to 11.87] | 1.542 [0.50 to 11.77]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non serious AEs were collected from the start of study treatment up to 196 days
Description: mITT population comprised of all randomized participants who were randomized apart from those randomized in error, received a treatment randomization number, modified and data for this population were based on actual treatment received. SAEs and AEs were reported for mITT Population.
Arm/Group | Placebo | Danirixin 5 mg | Danirixin 10 mg | Danirixin 25 mg | Danirixin 35 mg | Danirixin 50 mg
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102 | 1/103 | 2/103 | 1/102 | 1/102
Serious Adverse Events (participants affected / at risk) | 8/102 | 7/102 | 13/103 | 10/103 | 7/102 | 11/102
Other Adverse Events (participants affected / at risk) | 20/102 | 24/102 | 22/103 | 31/103 | 27/102 | 27/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Danirixin 5 mg (N=102) | Danirixin 10 mg (N=103) | Danirixin 25 mg (N=103) | Danirixin 35 mg (N=102) | Danirixin 50 mg (N=102)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Danirixin 5 mg (N=102) | Danirixin 10 mg (N=103) | Danirixin 25 mg (N=103) | Danirixin 35 mg (N=102) | Danirixin 50 mg (N=102)
Nasopharyngitis (Infections and infestations) | 12 (13) | 8 (8) | 9 (11) | 12 (14) | 14 (16) | 10 (14)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 7 (7) | 7 (8) | 9 (12) | 5 (8) | 6 (8)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 6 (6) | 5 (8) | 8 (9) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 4 (4) | 6 (7) | 5 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03034967/SAP_000.pdf
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03034967/Prot_001.pdf